CLINICAL TRIAL: NCT04729725
Title: Strategic Alliance: Phase 1b Trial Assessing Combination of TGF-β Inhibitor and PD-1 Inhibitor Cemiplimab
Brief Title: SAR439459 and Cemiplimab for the Treatment of Advanced or Unresectable Solid Tumors, Strategic Alliance, TACTIC TRIAL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The industry supporter discontinued the study and lead drug, SAR439459, due to toxicity.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0649; NCI-2020-10859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0649 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-11-30; First posted 2021-01-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SAR439459, cemiplimab) (Experimental): Patients receive SAR439459 IV over 30 minutes on day 1 and cemiplimab IV over 30 minutes on day 1 starting cycle 2. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-TGF-beta Monoclonal Antibody SAR-439459; Biological: Cemiplimab

INTERVENTIONS:
Biological: Anti-TGF-beta Monoclonal Antibody SAR-439459 — Given IV
  Other Names: Anti-TGFb SAR-439459; Anti-transforming Growth Factor-beta mAb SAR439459; SAR 439459; SAR-439459; SAR439459
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN2810

SUMMARY:
This is a phase Ib trial with SAR439459, a TGF-beta inhibitor, in combination with cemiplimab, a PD-L1 inhibitor, in patients with solid tumors that have spread to other places in the body (advanced) or cannot be removed by surgery (unresectable). Inhibiting TGF-beta may interfere with the ability of cancer cells to grow and spread and may sensitize cancers to immune checkpoint inhibitor therapy. The objective of this study is to determine whether this drug combination is effective in shrinking cancers, keeping them from growing, helping patients live longer, and to see if the drug combination is safe.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the anti-tumor activity of the combination of anti-TGF-beta monoclonal antibody SAR-439459 (SAR439459) and cemiplimab in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To confirm the safety and tolerability of the combination of SAR439459 and cemiplimab in patients with advanced solid tumors.

II. To evaluate the overall response rate (ORR), progression-free survival (PFS), median overall survival (OS) and duration of response (DoR).

III. To identify biomarkers of response and resistance to the combination of SAR439459 and cemiplimab in patients with advanced solid tumors.

OUTLINE:

Patients receive SAR439459 intravenously (IV) over 30 minutes on day 1 and cemiplimab IV over 30 minutes on day 1 starting cycle 2. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, and 90 days, then every 12 weeks until progression of disease is determined or patient receives additional anti-neoplastic medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed, advanced unresectable or metastatic solid tumor whom in the opinion of the Investigator do not have a suitable alternative therapy
* Disease must be measurable by Response Evaluation Criteria in Solid Tumors (RECIST 1.1), and safely undergo serial tumor biopsies. For patients with castration-resistant prostate cancer, evaluable disease by Prostate Cancer Working Group 3 (PCWG3) will be permitted if serial biopsies (e.g. bone tumor biopsies) are feasible
* Patients must have previously received a PD-1 or PD-L1 inhibitor-based therapy and must have achieved stable disease (SD) for at least 6 months, or complete remission/partial remission (CR/PR) prior to disease progression (secondary resistance) by radiological assessment by the study investigator. The PD-1 or PD-L1 inhibitor-based therapy must be the immediate line of treatment prior to study enrollment
* Patients must have adequate functional status as defined by Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000 / mcL
* Hemoglobin >= 9.0 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (creatinine clearance should be calculated per institutional standard)
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels >= 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Patients must have discontinued all previous systemic cancer treatments for at least 21 days and recovered from the acute toxic effects of therapy to grade < 1 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, excluding persistent grade 2 or higher toxicities determined to be clinically insignificant per the principal investigator (PI) (i.e. alopecia or grade 2 neuropathy). Patients must have discontinued from previous treatments as shown below:

  * Cytotoxic therapies or targeted agents that are small-molecule inhibitors >= 3 weeks prior to (study entry/enrollment/first dose of study treatment)
  * Mitomycin C or nitrosoureas >= 42 days prior to (study entry/enrollment/first dose of study treatment)
  * Biologic agents (e.g., antibodies) >= 3 weeks prior to (study entry/enrollment/first dose of study treatment)
  * Immunotherapy (e.g., CTLA4, PD-1, PDL1 inhibitors) >= 3 weeks prior to (study entry/enrollment/first dose of study treatment)
  * Radiotherapy >= 4 weeks prior to (study entry/enrollment/first dose of study treatment)
  * Limited field radiotherapy or palliative radiotherapy >= 3 weeks prior to (study entry/enrollment/first dose of study treatment)
  * Major surgery, excluding biopsy: Patients with recent major surgery must have recovered, in the opinion of the investigator, from the toxicity and/or complication from the intervention before starting therapy
  * Study drug with an investigational product, or non-approved use of a drug or device >= 3 weeks prior to (study entry/enrollment/first dose of study treatment)

    * If the patient was treated with an agent with a short half-life, washout can be < 3 weeks but no shorter than 5 times the half-life
* Women of child-bearing potential MUST have a negative serum or urine human chorionic gonadotropin (HCG) test at screening and within 2 days prior to receiving first dose of study treatment unless prior tubal ligation (>= 1 year before screening), total hysterectomy or menopause (defined as 12 consecutive months of amenorrhea). Patients should not become pregnant or breastfeed while on this study. Sexually active patients must agree to use dual contraception for the duration of study participation and for at least 6 months for females and 3 months for males after. Males should not donate sperm during the study and for 3 months after your last dose of study drugs
* Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients who have known active Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) infection
* Patients who have active infection requiring intravenous (IV) antibiotics or other uncontrolled intercurrent illness requiring hospitalization
* Patients unable to comply with the study and follow-up procedures
* Patients with history of cerebrovascular accident (CVA), myocardial infarction, clinically significant arrhythmia, unstable angina, pulmonary embolism, clinically significant deep vein thrombosis, gastrointestinal hemorrhage, clinically significant intestinal obstruction or perforation, or active uncontrolled bleeding within the previous 6 months before starting therapy
* Patients with a history of valvular heart disease (including valve replacement), known atrioventricular (A-V) malformation or evidence or history of septal aneurysm, other heart aneurysm, or any aneurysm of the major vessels
* Patients with a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Patients who have a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patients who have received a live vaccine within 30 days before the first dose of study treatment
* Patients who have symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids (patients receiving anticonvulsants are eligible)
* Patients who have primary central nervous system (CNS) tumors
* Patients with active known or suspected autoimmune disease or any illness that could compromise the immune system (e.g., prior organ transplant) within the past 2 years, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo, alopecia, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring chronic, and systemic immunosuppressive treatment within the past 2 years, not expected to recur in the absence of an external trigger, are permitted to enroll. Patients with inflammatory bowel disease and autoimmune related uveitis are not eligible
* Patients being treated with therapeutic doses of anticoagulants or antiplatelet agents (1 mg/kg of enoxaparin, 30 0mg of aspirin daily, 300 mg of clopidogrel daily or equivalent) within 7 days prior to first dose of SAR439459. Prophylactic use of anticoagulants or antiplatelets are allowed
* Prior treatment with any anti-transforming growth factor beta (TGFb) inhibitors
* Patients who received prior immunotherapy who developed toxicity leading to a permanent discontinuation of immunotherapy
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of SAR349459 and/or cemiplimab (occasional use of inhaled, intraocular, nasal or topical steroids for symptomatic relief allowed)
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, non-infectious pneumonitis that require immunosuppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in radiation field is permitted
* Prior history of CTCAE version 5.0 grade >= 1 or ongoing active uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | 12 weeks
  Defined as complete response (CR) + partial response (PR) + stable disease (SD) > 12 weeks > 12 weeks assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Will estimate CBR with 95% confidence intervals (CI). Will assess associations between marker levels and outcome using receiver operator characteristics curve analysis, graphical analysis and logistic regression analysis as appropriate.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 1 year after completion of study treatment
  AEs will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. AEs will be summarized by patient incidence rates, therefore, in any tabulation, a patient contributes only once to the count for a given AE preferred term. The number and percentage of patients with any treatment-emergent by NCI CTCAE v5.0 will be summarized for all study patients combined. The number and percentage of patients with treatment-emergent AEs assessed by the Investigator as at least possibly related to treatment will also be tabulated. The number and percentage of patients with any grade >= 3 treatment-emergent AE per NCI CTCAE v5.0 will be tabulated in the same manner. Serious AEs will also be tabulated.
Clinical benefit rate | Up to 1 year after completion of study treatment
  Defined as CR+PR+SD > 12 weeks assessed by immune-related (ir)RECIST. A 95% CI of response rate will be estimated based on the binomial distribution.
Overall response rate | Up to 1 year after completion of study treatment
  A 95% CI of response rate will be estimated based on the binomial distribution.
Progression free survival | Up to 1 year after completion of study treatment
  Will be summarized using Kaplan-Meier methodology using 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals, as well as percentage of censored observations.
Duration of response | Up to 1 year after completion of study treatment
  Assessed by RECIST v1.1 and irRECIST.
Overall survival | Up to 1 year after completion of study treatment
  Will be summarized using Kaplan-Meier methodology using 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals, as well as percentage of censored observations.
Correlation of somatic mutations | Up to 1 year after completion of study treatment
  Will be evaluated using whole-exome sequencing of pre-, on-treatment, and disease progression tumor biopsies. Will assess changes in frequency and type of mutations using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data.
Correlation of change in protein expression | Up to 1 year after completion of study
  Will be evaluated by reverse phase protein array (PPPA) analysis on pre-, on-treatment, and disease progression tumor biopsies. Will assess changes in normalized protein expression levels using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data.
Correlation of change in ribonucleic acid expression | Up to 1 year after completion of study
  Will be evaluated by ribonucleic acid (RNA) sequencing on pre-, on-treatment, and disease progression tumor biopsies. Will assess changes in normalized RNA expression levels using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data.
Circulating-free deoxynucleic acid as a biomarker of response and resistance | Up to 1 year after completion of study treatment
  Plasma for circulating-free deoxyribonucleic acid will be collected pre-, on-treatment, and at time of disease progression. Will assess changes in DN concentration levels using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data.
Peripheral mononuclear blood cells as a biomarker of response and resistance | Up to 1 year after completion of study treatment
  Peripheral mononuclear blood cells (PMBCs) from whole blood specimens will be collected pre-, on-treatment, and at time of disease progression. Will assess for changes in proportion of PMBC cell phenotypes using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data.
Cytokine levels as a biomarker of response and resistance | Up to 1 year after completion of study treatment
  Plasma for cytokine analysis will be collected pre-, on-treatment, and at time of disease progression. Will assess for changes in normalized cytokine levels using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data.
TGF-beta as a biomarker or response and resistance | Up to 1 year after completion of study treatment
  Plasma for TGF-beta analysis will be collected pre-, on-treatment, and at the time of disease progression. Will assess changes in normalized TGF-beta levels using paired t-tests for interval-scaled, normal data or Wilcoxon signed rank test for other numeric data, and exact version of McNemar's chi-squared test for binary data. Platelet factor 4 will be collected from plasma simultaneously as a marker of platelet contamination to monitor the quality of TGF-beta measurement.
Microbiome analysis | Baseline
  Fecal sample and buccal swab sample collected for 16S ribosomal RNA microbiome profiling analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Yap, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org